CLINICAL TRIAL: NCT06431204
Title: Obstetric Comorbidity Index for Prediction of Perioperative Severe Maternal Morbidity in Patients Undergoing Cesarean Delivery With Postpartum Hemorrhage
Brief Title: Obstetric Comorbidity Index in Postpartum Hemorrhage
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 351/2567(IRB2); Si 359/2024 (Other: Siriraj Institutional Review Board)
Record Dates: First submitted 2024-05-17; First posted 2024-05-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section Complications; Postpartum Hemorrhage; Morbidity;Perinatal
Keywords: cesarean section; postpartum hemorrhage; maternal morbidity; obstetrics comorbidity index
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with postpartum hemorrhage with severe maternal morbidity: Patients with either one of severe maternal morbidity (severe hemorrhage, hypertension/neurologic, renal, sepsis, pulmonary, cardiac, intensive care unit, and anesthesia complications)
  Interventions: Other: Obstetric comorbidity index
- Patients with postpartum hemorrhage without severe maternal morbidity: Patients without the severe maternal morbidity conditions
  Interventions: Other: Obstetric comorbidity index

INTERVENTIONS:
Other: Obstetric comorbidity index — Obstetric comorbidity index score

SUMMARY:
The objective of this study is to examine the predictive capability of the Obstetric comorbidity index in the identification of severe maternal morbidity associated with postpartum hemorrhage in patients undergoing cesarean delivery.

DETAILED DESCRIPTION:
The prospectively predictive maternal morbidity is imperative to enhance maternal outcomes. There has been development of the obstetric comorbidity index (OBCMI) by Bateman et al. in 2013 and performed with superior performance characteristics relative to general comorbidity measures in an obstetric population. The score has been a growing recognition of the necessity for specialized risk assessment tools tailored specifically to obstetric populations that differ from other populations. For instance, both the Charlson/Romano comorbidity index or the Elixhauser comorbidity score and their adaptations are deficient in accounting for obstetric conditions, thereby limiting their ability to predict obstetric morbidity or mortality.

The Obstetric Comorbidity Index has undergone thorough examination and validation across multiple nations. These findings collectively demonstrate the index's capacity for moderate to high predictive accuracy in anticipating maternal morbidities, accompanied by a commendable discriminative performance.

However, within the context of Thailand, investigations concerning the Obstetric Comorbidity Index and its association with perioperative complications or morbidities in postpartum hemorrhage patients undergoing cesarean delivery remain unexplored. Therefore, this study aims to elucidate the correlation between the Obstetric Comorbidity Index and severe maternal morbidity, while also scrutinizing the prevalence of comorbidities during the perioperative period among patients undergoing cesarean delivery at the largest University hospital, in THAILAND. Predicting the rate of maternal morbidity would be advantageous for facilitating preparation and augmenting awareness of complications during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

The patients underwent cesarean delivery with the diagnosis of postpartum hemorrhage (ICD-10 coding O72.1)

Exclusion Criteria:

* Cesarean delivery at less than 24 weeks of gestation
* A patient chart that does not contain primary outcome data eg. absence of anesthetic record
* Blood loss less than 1,000 ml in the first 24 hours postpartum

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The chart of patients who underwent cesarean delivery with the diagnosis of postpartum hemorrhage (bleeding >, = 1,000 ml) and gestational age of more than 24 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2024-07-13 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
The prediction of severe maternal morbidity using obstetric comorbidity index | in 72 hours after cesarean delivery
  The prediction of severe maternal morbidity using obstetric comorbidity index presented in C-statistic (AUC of ROC)

SECONDARY OUTCOMES:
Rate of blood transfusion | in 72 hours after cesarean delivery
  Perioperative red blood cells transfusion in units
Quantity of postpartum hemorrhage | in 24 hours after cesarean delivery
  Quantity of postpartum hemorrhage in ml.
Cause of postpartum hemorrhage | in 24 hours after cesarean delivery
  Main cause of postpartum hemorrhage
Rate of ICU admission | in 24 hours after cesarean delivery
  Rate of intensive care unit admission
Rate of Postoperative complications | in 72 hours after cesarean delivery
  Post operative complications eg. congestive heart failure, TRALI, acute kidney injury
Neonatal Apgar score | at 1-minute and 5-minute after delivery
  Neonatal Apgar score from 0 - 10
Rate of maternal mortality | in 72 hours after cesarean delivery
  Maternal death rate

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok THAILAND
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
The investigators may balance the potential benefits and risks for each request and then provide the data that could be shared, together with the permission from the hospital director.